CLINICAL TRIAL: NCT04406675
Title: Social Cognition in Patients With Amyotrophic Lateral Sclerosis
Acronym: COSISLA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020-A01213-36
Record Dates: First submitted 2020-05-13; First posted 2020-05-28 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-06

CONDITIONS: Social Cognition
MeSH Terms: interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients Amyotrophic Lateral Sclerosis (Other)
  Interventions: Other: neuropsychological test
- Control subjects (Other)
  Interventions: Other: neuropsychological test

INTERVENTIONS:
Other: neuropsychological test — neuropsychological test

SUMMARY:
Amyotrophic Lateral Sclerosis, also known as Charcot disease, is a neurodegenerative disease evidenced by gradual paralysis of the muscles involved in voluntary motor function. The clinical hallmark of Amyotrophic Lateral Sclerosis is the combination of upper and lower motor neuron signs and symptoms. The most recent studies suggest that up to 50% of Amyotrophic Lateral Sclerosis patients demonstrate mild to moderate cognitive disturbance. Impaired social cognition, including a deficit in the recognition of facial emotions and the identification of vocal prosody, is recognized as a part of the cognitive phenotype of Amyotrophic Lateral Sclerosis, with crucial implications for patients' and caregivers' training. However, studies remain scarce and the data acquired must be supported. The evolution of these manifestations during the disease is still poorly understood.

In this study the investigators aim to assess the social cognition capacities of patients with Amyotrophic Lateral Sclerosis compared to healthy matched control subjects.

ELIGIBILITY:
Inclusion Criteria:

Patient Amyotrophic Lateral Sclerosis :

* Education of at least 7 years
* Native language: French
* Patients Amyotrophic Lateral Sclerosis
* Signature of informed consent to participate in the study
* Accompanied patient

Control subject :

* People without any pathology
* Education of at least 7 years
* Native language: French
* Signature of informed consent to participate in the study

Exclusion Criteria:

Patient Amyotrophic Lateral Sclerosis and control subject :

* Simultaneous participation in another interventional protocol with experimental treatment
* Inability to perform cognitive study tests
* Pregnant, lactating or parturient women
* Persons deprived of their liberty by administrative or judicial decision
* Persons under psychiatric care under duress
* Persons subject to legal protection measures
* Persons out of state to express their consent
* People not affiliated or not beneficiaries of a social security scheme
* History likely to disturb cognition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2020-09-21 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Evaluate the social cognition capacities | One day
  Evaluate the social cognition capacities of patients with Amyotrophic Lateral Sclerosis compared to control subjects using dynamic social cognition tests : Movie for the Assessment of Social Cognition. The maximum score is 48 points. The higher the score for correct answers, the better the performance.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Angers, Angers, France

REFERENCES:
- [Derived] Faure-de Baets J, Besnard J, Cassereau J, Emmelin E, Allain P. Assessment of social cognition in patients with amyotrophic lateral sclerosis: protocol for a cross-sectional comparative study at Angers University Hospita. BMJ Open. 2025 Jul 5;15(7):e097543. doi: 10.1136/bmjopen-2024-097543. PMID 40617623